CLINICAL TRIAL: NCT04914728
Title: Mini-invasive Lumbar Arthrodesis in Ambulatory: Pilot Study "ALAMBU"
Brief Title: Mini-invasive Lumbar Arthrodesis in Ambulatory
Acronym: ALAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALAMBU; 2020-A01211-38 (Other: ANSM)
Record Dates: First submitted 2021-05-17; First posted 2021-06-07 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Lumbar Spine Degeneration
Keywords: mini-invasive lumbar arthrodesis

STUDY DESIGN:
Intervention Model Description: Single-centre, pilot study evaluating the feasibility, difficulties and morbidity of ambulatory lumbar arthrodesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mini-invasive lumbar arthrodesis (Experimental): The patient will be admitted to the hospital on the morning of the surgery, operated on the same morning by either the posterior or anterior mini-invasive approach.
  The choice of the approach depends on the specificity of the pathology leading to the arthrodesis procedure and the surgeon's experience. It is the surgeon who decides this in agreement with the patient. The patient will be discharged in the evening after agreement of the anaesthetist and the surgeon.
  Interventions: Procedure: mini-invasive lumbar arthrodesis

INTERVENTIONS:
Procedure: mini-invasive lumbar arthrodesis — * The mini-invasive posterior approach is performed using a trans-muscular Wiltse approach. Pedicle screws, neurological decompression and intersomatic cage placement are performed.
  * The mini-invasive anterior approach is performed via a left retroperitoneal pararectal approach. After complete discectomy, an intersomatic cage stabilised by a screwed plate will be placed.

SUMMARY:
Degenerative lumbar pathologies are characterised by functional impairment and the occurrence of severe chronic pain and disability Arthrodesis of the lumbar spine is a common surgery for the treatment of degenerative lumbar pathologies. It is commonly performed during a hospital stay that can vary from 3 to 7 days. The development of mini-invasive techniques and the development of the Improved Rehabilitation after Surgery programmes, has considerably reduced the hospital stay of the patients. It is possible that in the future mini-invasive lumbar arthrodesis will be performed on an ambulatory as a standard procedure, but its safety, efficacy and patient satisfaction must be proven and validated.

DETAILED DESCRIPTION:
Degenerative lumbar disease (DLD) is a condition of increasing frequency, affecting millions of patients worldwide. They are characterised by functional impairment and the occurrence of severe chronic pain and disability.

Arthrodesis of the lumbar spine is a common surgery for the treatment of DLD. It is commonly performed during a hospital stay that can vary from 3 to 7 days. The advent of mini-invasive techniques and the development of Improved Rehabilitation after Surgery program has made it possible to considerably reduce the duration of hospitalization of patients with a high rate of satisfaction, a reduction in costs and without increasing morbidity. In spinal surgery, decompression procedures such as discectomy and lumbar recalibration are frequently performed on an ambulatory. The first American studies with a low level of evidence on the management of mini-invasive lumbar arthrodesis are beginning to appear. It is quite possible that in the future this type of procedure will be carried out on an ambulatory as a standard procedure, but its safety, efficacy and patient satisfaction must be proven and validated. In the United States, 23-hour hospitalizations are considered as ambulatory procedures, whereas in France, ambulatory is qualified as such when the patient is admitted and discharged in the same day.

The study population was patients who had failed medical treatment (analgesics and rehabilitation) for more than three months and who required a mono-segmental arthrodesis procedure for the management of their lumbar-radiculalgia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Patients affiliated to a social security system.
* Informed, dated and signed consent
* ASA 1 or 2
* Patient compliant and adhering to protocol visits
* Indication for a 1-level mini-invasive lumbar arthrodesis performed by anterior or posterior approach
* Failure of conservative treatment for more than 3 months

Exclusion Criteria:

* History of lumbar arthrodesis
* Active neoplasia
* History of osteoporotic fractures of the spine
* Arthrodesis superior to 1 level
* Intolerance or contraindication to morphine treatments
* Respiratory insufficiency
* Preoperative anticoagulant treatment
* Contraindication to the ambulatory care: patient living alone at home, or at a distance from the establishment, and thus requiring a follow-up care and rehabilitation hospitalization
* Patient with a body mass index of greater than 40 kg/m².
* Patient with a fever (>38°C)
* Suspected or known allergy or intolerance to the materials used and requiring a combination of different metals.
* Patient with a contraindication to the material used or for whom the use of the implant could interfere with their anatomical structures or expected physiological function.
* Pregnant or breastfeeding women
* Patient participating to an ongoing study that may interfere with the present study
* Patient under legal protection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility of mini-invasive lumbar arthrodesis on an ambulatory in patients with degenerative lumbar disease who have failed with conventional treatment. | within 24 hours after surgery
  Percentage of patients with same-day discharge

SECONDARY OUTCOMES:
Evaluate the safety of ambulatory lumbar arthrodesis | through study completion, an average of 1 year
  Record of adverse event
Evaluate early morbidity | within 1st week
  Occurrence of re-hospitalization and/or emergency readmission and/or need for re-operation of the patient
Evaluate the short-term morbidity | within 1st month
  Presence of a cicatrization disorder, the occurrence of an infection, neurological damage, adverse event related to the implants, vascular and/or medical problem.
Evaluate the mid-term morbidity | within 1st year
  occurrence of pseudoarthrosis
Evaluate the patients' quality of life | at 1-month visit
  Short Form-36 Health Survey questionnaire
Evaluate the patients' quality of life | at 1-month visit
  Evaluated by Oswestry
Evaluate the patients' quality of life | at 6-month visit
  Evaluated by Short Form-36 Health Survey questionnaire
Evaluate the patients' quality of life | at 6-month visit
  Evaluated by Oswestry
Evaluate the patients' quality of life | at 1-year visit
  Evaluated by Short Form-36 Health Survey questionnaire
Evaluate the patients' quality of life | at 1-year visit
  Evaluated by Oswestry
Evaluate the patients' quality of life | at 1-month visit
  Return to professional activity
Evaluate the patients' quality of life | at 6-month visit
  Return to professional activity
Evaluate the patients' quality of life | at 1-year visit
  Return to professional activity
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: L1S1 lumbar lordosis
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: Segmental lordosis of the arthrodesis level
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: Pelvic Incidence
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: Pelvic version
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: Sacral slope
Evaluate radiological parameters | at 1-month visit
  The radiological parameter: Disc height
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: L1S1 lumbar lordosis
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: Segmental lordosis of the arthrodesis level
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: Pelvic Incidence
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: Pelvic version
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: Sacral slope
Evaluate radiological parameters | at 6-month visit
  The radiological parameter: Disc height
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: L1S1 lumbar lordosis
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: Segmental lordosis of the arthrodesis level
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: Pelvic Incidence
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: Pelvic version
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: Sacral slope
Evaluate radiological parameters | at 1-year visit
  The radiological parameter: Disc height
Evaluate patient satisfaction with the procedure | at 1-month visit
  Satisfaction score
Evaluate patient satisfaction with the procedure | at 6-month visit
  Satisfaction score
Evaluate patient satisfaction with the procedure | at 1-year visit
  Satisfaction score
Evaluate lumbar pain | at 1-month visit
  Lumbar Visual Analogue Scales pain
Evaluate lumbar pain | at 6-month visit
  Lumbar Visual Analogue Scales pain
Evaluate lumbar pain | at 1-year visit
  Lumbar Visual Analogue Scales pain
Evaluate radicular pain | at 1-month visit
  Radicular Visual Analogue Scales pain
Evaluate radicular pain | at 6-month visit
  Radicular Visual Analogue Scales pain
Evaluate radicular pain | at 1-year visit
  Radicular Visual Analogue Scales pain
Evaluate lumbar and radicular pain | before the 1-month visit
  record of analgesic treatments taken before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Louis BOISSIERE, MD, Principal Investigator — Unité de Chirurgie de la Colonne Vertébrale
Locations (1):
- Unité de Chirurgie de la Colonne Vertébrale, Bruges, France

REFERENCES:
- [Background] Hoy D, Brooks P, Blyth F, Buchbinder R. The Epidemiology of low back pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):769-81. doi: 10.1016/j.berh.2010.10.002. PMID 21665125
- [Background] Peng CW, Yue WM, Poh SY, Yeo W, Tan SB. Clinical and radiological outcomes of minimally invasive versus open transforaminal lumbar interbody fusion. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1385-9. doi: 10.1097/BRS.0b013e3181a4e3be. PMID 19478658
- [Background] Dietz N, Sharma M, Adams S, Alhourani A, Ugiliweneza B, Wang D, Nuno M, Drazin D, Boakye M. Enhanced Recovery After Surgery (ERAS) for Spine Surgery: A Systematic Review. World Neurosurg. 2019 Oct;130:415-426. doi: 10.1016/j.wneu.2019.06.181. Epub 2019 Jul 2. PMID 31276851
- [Background] Sivaganesan A, Hirsch B, Phillips FM, McGirt MJ. Spine Surgery in the Ambulatory Surgery Center Setting: Value-Based Advancement or Safety Liability? Neurosurgery. 2018 Aug 1;83(2):159-165. doi: 10.1093/neuros/nyy057. PMID 29538716
- [Background] Wiltse LL, Bateman JG, Hutchinson RH, Nelson WE. The paraspinal sacrospinalis-splitting approach to the lumbar spine. J Bone Joint Surg Am. 1968 Jul;50(5):919-26. No abstract available. PMID 5676831
- [Background] Harmon PH. A simplified surgical technic for anterior lumbar diskectomy and fusion; avoidance of complications; anatomy of the retroperitoneal veins. Clin Orthop Relat Res. 1964 Nov-Dec;37:130-44. No abstract available. PMID 5889125
- [Background] Perneger TV, Leplege A, Etter JF, Rougemont A. Validation of a French-language version of the MOS 36-Item Short Form Health Survey (SF-36) in young healthy adults. J Clin Epidemiol. 1995 Aug;48(8):1051-60. doi: 10.1016/0895-4356(94)00227-h. PMID 7775992
- [Background] Hayashi K, Boissiere L, Guevara-Villazon F, Larrieu D, Nunez-Pereira S, Bourghli A, Gille O, Vital JM, Pellise F, Sanchez Perez-Grueso FJ, Kleinstuck F, Acaroglu E, Alanay A, Obeid I. Factors influencing patient satisfaction after adult scoliosis and spinal deformity surgery. J Neurosurg Spine. 2019 May 10;31(3):408-417. doi: 10.3171/2019.2.SPINE181486. Print 2019 Sep 1. PMID 31075761
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476